CLINICAL TRIAL: NCT04379310
Title: Evaluation of Demographic and Clinical Parameters on Admission and Medications Used for Comorbidities in Patients With Covid-19 Pneumonia: A Single Center Experience in Turkey
Brief Title: Evaluation of Clinical Parameters on Admission and Medications in Covid-19 Pneumonia (Corona Virus Disease 2019)
Acronym: Covid-19
Status: Completed | Type: Observational
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Murat Civan, M.D., Istanbul Nisantasi University
Other Study IDs: 20200504441
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Covid-19
Keywords: covid-19 pneumonia; medication; comorbidity
MeSH Terms: conditions — COVID-19 | interventions — Angiotensin-Converting Enzyme Inhibitors; Calcium Channel Blockers; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid-19 pneumonia: diagnosed with covid-19 by using PCR and computed tomography scans
  Interventions: Drug: ACE Inhibitors and Calcium Channel Blockers

INTERVENTIONS:
Drug: ACE Inhibitors and Calcium Channel Blockers — effect of drugs on patients with covid-19 pneumonia
  Other Names: NSAID

SUMMARY:
Investigators will recruit patients diagnosed with COVID-19 pneumonia between March 11th, 2020 and April 15th, 2020 in emergency, internal medicine and cardiology outpatient clinics, retrospectively and analyze their clinical and demographic features on admission in regard to their medications used for chronic diseases regularly.

DETAILED DESCRIPTION:
Covid-19 infections demonstrated a pandemic spread after January 2020 and their associations with patient characteristics and comorbidities are intensely studied. Investigators also want to find out potential relations between major medications taken for chronic diseases and clinical parameters of patients with Covid-19 pneumonia.

For the study, investigators will recruit patients diagnosed with COVID-19 pneumonia between March 11th, 2020 (the date at which the first case of Covid-19 in Turkey officially declared) and April 15th, 2020 in emergency, internal medicine and cardiology outpatient clinics, retrospectively. All of the demographic features, complaints on admission, reports of computed tomography (CT) scans of the chest without intravenous contrast issued by the staff radiologist, c-reactive protein (CRP) and complete blood count (CBC) values on admission will be recorded retrospectively. Their polymerase chain reaction (PCR) test results will be derived from the hospital records based on public health covid-19 database notifications and list of medications taken regularly for more than 8 weeks before the diagnosis of COVID-19 pneumonia from the national pharmacy database. Information about other systemic diseases and major medical conditions of patients will be procured from the medical histories gained by relevant physicians. Patient taking each drug group will be compared to those not taking that drugs in terms of clinical and demographical features mentioned above. Statistical analysis will be performed by using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 pneumonia at least with typical infiltration on CT +/- positive PCR.

Exclusion Criteria:

* no typical infiltration and negative PCR results.
* not newly diagnosed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: first diagnosis with covid-19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
extend of lung involvement | 1 week
  number of segments involved on admission
oxygen saturation on admission | 2 week
  hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Haciosman, Study Chair — academic staff, MD
Locations (1):
- Vital Hospital, Bahçelievler, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
patient characteristics and time interval will be shared
Supporting Information: Study Protocol
Time Frame: in two months
Access Criteria: all researchers